CLINICAL TRIAL: NCT01000090
Title: Surgical Versus Medical Treatment of Acromegaly: Effects on Biochemical Markers
Brief Title: Surgical Versus Medical Treatment of Acromegaly
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: kzr200809
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2011-06

CONDITIONS: Acromegaly
Keywords: Acromegaly; Somatostatin analogues; Treatment
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acromegaly patients, somatostain analogues
- Acromegaly patients, surgery

SUMMARY:
Evaluate biochemical differences in acromegalic patients treated with surgery versus somatostatin analogues (SMS) (after surgery or alone).

Hypothesis: Treatment modality exhibit different biochemical responses in acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Acromegaly diagnosis
* treated with Somatostatin analogues or surgery
* in treatment control

Exclusion Criteria:

* treatment with GH-antagonist
* never treated
* not in treatment control

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acromegalic patients followed in the outpatient clinic at Århus University Hospital, Medical Department M
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Z Rubeck, stud. med., Study Director — Medical department M, Århus University Hospital; Jens Otto L Jørgensen, MD, Principal Investigator — Medical department M, Århus University Hospital; Michael Madsen, MD, Study Director — Medical department M, Århus University Hospital; Sanne Fisker, MD, Study Director — Medical department M, Århus University Hospital; Caroline Adreasen, MD, Study Director — Medical department M, Århus University Hospital; Jan Frystyk, MD, Study Director — Medical department M, Århus University Hospital
Locations (1):
- Århus University Hospital, Medical department M, Aarhus, Denmark